CLINICAL TRIAL: NCT00758784
Title: Safety and Efficacy of an Ophthalmic Solution in Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-S&E-0417082-P
Record Dates: First submitted 2008-09-19; First posted 2008-09-25 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bromfenac ophthalmic solution 0.06% (Experimental): bromfenac ophthalmic solution 0.06% bilaterally twice a day
  Interventions: Drug: bromfenac ophthalmic solution 0.06%

INTERVENTIONS:
Drug: bromfenac ophthalmic solution 0.06% — bromfenac ophthalmic solution 0.06% bilaterally twice a day

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of an ophthalmic solution in dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older

Exclusion Criteria:

* No active ocular conditions of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-08-13; Primary Completion 2009-01-14 (Actual); Study Completion 2009-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
Started | 38
Completed | 36
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Average Lissamine Green Staining in the Study Eye
Description: Lissamine green staining was assessed for both eyes at each study visit. The Investigator inserted a lissamine green staining strip into the inferior conjunctival cul-de-sac. Staining density for each of the 6 regions of the conjunctiva (temporal, superior temporal, inferior temporal, superior nasal, inferior nasal, and nasal) was graded from 0 to 3 approximately 2.5 minutes after strip instillation according to the National Eye Institute (NEI) chart and grid. The scale for total scoring ranged from 0 to 18 units summed across all 6 conjunctival regions, with a higher score suggesting a more dry eye condition. An average of the 6 areas was computed, providing an average score of 0-3 units. The study eye utilized for analysis was selected by pre-specified criteria.
Time Frame: Baseline, Day 42
Population: All participants enrolled were included in the analysis population, with last observation carried forward applied for missing values.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
Number analyzed (Participants) | 38
score on a scale | -0.65 (0.40)

2. Primary Outcome: Percentage of Participants With at Least One Adverse Event
Time Frame: 52 days
Measure: Count of Participants; unit: Participants
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
Number analyzed (Participants) | 38
Participants | 9

3. Secondary Outcome: Mean Change From Baseline to Worst Region in Lissamine Green Staining in the Study Eye
Description: Lissamine green staining was assessed for both eyes at each study visit. The Investigator inserted a lissamine green staining strip into the inferior conjunctival cul-de-sac. Staining density for each of the 6 regions of the conjunctiva (temporal, superior temporal, inferior temporal, superior nasal, inferior nasal, and nasal) was graded from 0 to 3 approximately 2.5 minutes after strip instillation according to the National Eye Institute (NEI) chart and grid. The scale for worst region of Lissamine Green staining ranged from 0 to 3 units, with a higher score suggesting a more dry eye condition.The worst region of lissamine green staining was determined at the baseline visit. The study eye utilized for analysis was selected based on pre-specified criteria.
Time Frame: Baseline, 42 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
Number analyzed (Participants) | 38
score on a scale | -0.84 (0.75)

ADVERSE EVENTS:
Time Frame: 52 days
Arm/Group | Bromfenac Ophthalmic Solution 0.06%
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Ophthalmic Solution 0.06% (N=38)
Nasopharyngitis (Infections and infestations) | 2

LIMITATIONS AND CAVEATS:
Participants could co-administer Refresh Plus OTC eyedrops as needed during treatment/follow-up. Only 29 participants dosed all 42 days. Environmental factors influencing dry eye (eg, temperature, humidity, season, geography) were not controlled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.